CLINICAL TRIAL: NCT05498675
Title: Effect of Sacubitril/Valsartan on Cardiac Function Assessed by Cardiac Magnetic Resonance (CMR) in Hypertensive Patients Stratified by Body Mass Index (BMI): A Real World Study
Brief Title: Effect of Sacubitril/Valsartan on Cardiac Function in Hypertensive Patients Stratified by BMI: A Real World Study
Status: Recruiting | Type: Observational
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2022-P2-173-01
Record Dates: First submitted 2022-08-01; First posted 2022-08-12 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Sacubitril/Valsartan; Hypertension; Obesity
Keywords: Cardiac function; Cardiac magnetic resonance
MeSH Terms: conditions — Hypertension; Obesity | interventions — sacubitril; Valsartan; sacubitril and valsartan sodium hydrate drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Sacubitril/valsartan group: Patients administered sacubitril / valsartan oral tablet (Entresto) 200mg 1/day by prescription that have started before inclusion of the patient enrolled into the study and defined as sacubitril/valsartan group.
  Interventions: Drug: Sacubitril / Valsartan Oral Tablet [Entresto]
- ACEI/ARB group: Patients administered angiotensin-converting enzyme inhibitors/angiotensin II receptor antagonists (ACEI/ARB) by prescription that have started before inclusion of the patient enrolled into the study and defined as ACEI/ARB group.
  Including:
  benazepril, captopril, enalapril, fosinopril, lisinopril, moexipril, perindopril, quinapril, ramipril, trandolapril, azilsartan, candesartan, eprosartan, irbesartan, losartan, olmesartan, telmisartan, valsartan.
  Interventions: Drug: ACEI/ARB

INTERVENTIONS:
Drug: Sacubitril / Valsartan Oral Tablet [Entresto] — There is no treatment allocation. Patients administered sacubitril / valsartan oral tablet (Entresto) 200mg 1/day by prescription that have started before inclusion of the patient enrolled into the study and defined as sacubitril/valsartan group.
  Groups: Sacubitril/valsartan group
Drug: ACEI/ARB — There is no treatment allocation. Patients administered angiotensin-converting enzyme inhibitors/angiotensin II receptor antagonists (ACEI/ARB) by prescription that have started before inclusion of the patient enrolled into the study and defined as ACEI/ARB group.
  Including:
  benazepril, captopril, enalapril, fosinopril, lisinopril, moexipril, perindopril, quinapril, ramipril, trandolapril, azilsartan, candesartan, eprosartan, irbesartan, losartan, olmesartan, telmisartan, valsartan.
  Groups: ACEI/ARB group

SUMMARY:
The purpose of this study is to investigate the effect of sacubitril/valsartan on cardiac function assessed by cardiac magnetic resonance (CMR) in hypertensive patients stratified by BMI.

DETAILED DESCRIPTION:
Obesity is one of the risk factors of hypertension, and affects cardiac structure and function in the long term for hypertensive patients. Sacubitril/valsartan is regarded as a better antihypertensive drug for the improvement of cardiac function for patients with heart failure, but it remains unclear whether there are differences among different BMI groups. Therefore, the aim of this study was to evaluate the benefit of sacubitril/valsartan versus other antihypertensive drugs on cardiac structure and function assessed by CMR in hypertensive patients stratified by BMI in the real world.

ELIGIBILITY:
Inclusion Criteria:

* Patients with essential hypertension
* 18-70 years old
* No major barriers to provide written consent

Exclusion Criteria:

* Secondary hypertension, except because of sleep apnea
* cardiovascular disease (myocardial infarction, heart failure, stroke or coronary revascularization) within 6 months
* Severe concomitant diseases (autoimmune disease, malignancy, late stage of liver diseases, respiratory diseases and digestive diseases)
* Unable to understand or comply with the study procedures

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hypertensive patients stratified by BMI.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes on left ventricular ejection fraction (LVEF) | 6 months
  Changes on LVEF in % assessed with the use of cardiac magnetic resonance (CMR).

SECONDARY OUTCOMES:
Changes on left ventricular end-systolic diameter (LVESD) | 6 months
  Changes on LVESD in mm assessed with the use of CMR.
Changes on left ventricular end-diastolic diameter (LVEDD) | 6 months
  Changes on LVEDD in mm assessed with the use of CMR.
Changes on cardiac systolic function | 6 months
  Changes on cardiac systolic function in E/A, E-wave deceleration time (EDT) in ms assessed with the use of CMR.
Major adverse cardiac events | 6 months
  Including all-cause mortality, cardiac death, acute myocardial infarction, stroke, heart failure, ventricular tachycardia or ventricular fibrillation requiring shock delivery.
Major adverse cardiac events | 12 months
  Including all-cause mortality, cardiac death, acute myocardial infarction, stroke, heart failure, ventricular tachycardia or ventricular fibrillation requiring shock delivery.
Changes on hypertension-mediated target organ damage | 12 months
  Change on hypertension-mediated target organ damage including the estimated glomerular filtration rate (eGFR), total cholesterol, triglycerides level, LDL-cholesterol, HDL-cholesterol, and carotid intima-media thickness (IMT) assessed by carotid ultrasound
Changes on blood pressure | 6 months
  Changes on systolic and blood pressure assessed with the use of 24-hour ambulatory blood pressure monitoring (ABPM).
Changes on blood pressure | 12 months
  Changes on systolic and blood pressure assessed with the use of 24-hour ABPM.

CONTACTS AND LOCATIONS:
Overall Officials: Rongchong Huang, M.D., Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No